CLINICAL TRIAL: NCT02414711
Title: Validation of the French Translation of the Scale HSCL25 in the Diagnosis of Depression in Primary Care
Acronym: HSCL25
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HSCL25 Validation
Record Dates: First submitted 2015-03-19; First posted 2015-04-13 (Estimated); Last update posted 2025-12-03 (Actual); Status verified 2017-01

CONDITIONS: Depression
Keywords: Depression; Primary care; General Practitioners
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No depressed (Other): If the result of the HSCL25 scale is inferior than 1.75, then the patient is considered as no depressed.
  50 of these patients have to have a psychological interview with the PSE9 questionary to validate the result of the HSCL25 scale.
  Interventions: Other: HSCL25 scale; Other: PSE9 questionary
- Depressed (Other): If the result of the HSCL25 scale is superior or equal to 1.75, then the patient is considered as depressed.
  50 of these patients have to have a psychological interview with the PSE9 questionary to validate the result of the HSCL25 scale.
  Interventions: Other: HSCL25 scale; Other: PSE9 questionary

INTERVENTIONS:
Other: HSCL25 scale — The patient must answer to 25 questions of the HSCL25 scale. In function of the results, the patients was diagnosed depressed (≥1.75) or not depressed (<1.75)
Other: PSE9 questionary — On the 900 patients recruited, 50 patients who was diagnosed depressed or no depressed have to have a psychological interview with the PSE9 questionary to validate the first diagnosis done by the HSCL25 scale

SUMMARY:
Depression has emotional consequences, social and important business. Reaching at least 7.5% of French aged 15 to 85 years. General Practitioners are the first professional consulted in terms of frequency of consultations. Indeed, in primary care, 10 to 25% of patients with depression that General Practitioners are often alone to support and follow. But General Practitioners are faced with diagnostic difficulties facing the diagnosis of depression, because if the patient does not engage itself, no tool is validated in France to help them in their diagnosis. However, standardized questionary exist that allow to overcome this difficulty. Questionary used in other european countries. Among them, the HSCL25 scale was selected by a systematic review of literature and a RAND UCLA type of consensus procedure. This HSCL25 scale is the most efficient for the diagnosis of depression in terms of efficiency tool, reproducibility and ergonomics. However, it remains necessary to confirm its validity in terms of the French translation and in terms of efficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 and over) consultant in primary care

Exclusion Criteria:

* Child or young person under 18
* Women with a declared pregnancy to prevent puerperal depression whose support is different.
* Adult consultant to obtain a medical certificate
* Psychotic patients and\or requiring immediate care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1128 (Actual)
Dates: Start 2015-06; Primary Completion 2016-02 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
To validate the French translation of the HSCL25 scale | 1 month
  The score between HSCL25 scale and PSE9 questionary will be compared
To assess the HSCL25 scale diagnosis efficacy of depression in primary care ambulatory practice | 1 month
  The score between HSCL25 scale and PSE9 questionary will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Patrice NABBE, GP, Principal Investigator — GP department
Locations (3):
- France (3):
  - Cabinet médical en zone urbaine, Brest, France
  - Cabinet médical en zone rurale - Pôle Santé Universitaire, Lanmeur, France
  - Cabinet médical en zone semi-rurale, Plounéour-Trez, France

REFERENCES:
- [Result] Nabbe P, Le Reste JY, Guillou-Landreat M, Gatineau F, Le Floch B, Montier T, Van Marwijk H, Van Royen P. The French version of the HSCL-25 has now been validated for use in primary care. PLoS One. 2019 Apr 4;14(4):e0214804. doi: 10.1371/journal.pone.0214804. eCollection 2019. PMID 30946774